CLINICAL TRIAL: NCT06846606
Title: A Phase 1 Study of AUTX-703 in Participants With Relapsed/Refractory Acute Myeloid Leukemia and Myelodysplastic Syndromes
Brief Title: Phase 1 Study of AUTX-703 in Relapsed/Refractory AML and MDS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Auron Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AUTX-703-001
Record Dates: First submitted 2025-02-06; First posted 2025-02-26 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Relapsed Acute Myeloid Leukemia (AML); Refractory Acute Myeloid Leukemia (AML); Relapsed/Refractory AML; Relapsed Myelodysplastic Syndromes; Refractory Myelodysplastic Syndromes; Relapsed/Refractory (R/R) Acute Myeloid Leukemia (AML)
Keywords: AUTX-703; Relapsed Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia; Relapsed/Refractory AML; Acute Myeloid Leukemia; Relapsed Myelodysplastic Syndromes; Refractory Myelodysplastic Syndromes; KAT2A/B degrader; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Recurrence

STUDY DESIGN:
Intervention Model Description: This study consists of two parts: Part A (Dose Escalation) and Part B (Dose Optimization). In Part A, participants are assigned sequentially to escalating dosages of AUTX-703 to determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D). In Part B, participants are randomly assigned to receive one of two dosages of AUTX-703 for safety, pharmacokinetics, pharmacodynamics, and preliminary clinical activity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation - Part A (Experimental): Participants will receive escalating dosages of AUTX-703 orally in tablet form once, twice or three times weekly to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D).
  Interventions: Drug: AUTX-703
- Dose Optimization - Part B, Dosage 1 (Experimental): Participants will receive AUTX-703 at the first selected dosage determined from Part A, administered orally in tablet form either once, twice or three times weekly to further evaluate safety, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity at this specified dose.
  Interventions: Drug: AUTX-703
- Dose Optimization - Part B, Dosage 2 (Experimental): Participants will receive AUTX-703 at the second selected dosage determined from Part A, administered orally in tablet form either once, twice or three times weekly to further evaluate safety, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity at this specified dose.
  Interventions: Drug: AUTX-703

INTERVENTIONS:
Drug: AUTX-703 — AUTX-703 administered orally

SUMMARY:
This Phase 1, multicenter, open-label, dose escalation and dose optimization study is designed to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity of AUTX-703 administered orally in subjects with advanced hematologic malignancies.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1, multicenter study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity of AUTX-703, an orally bioavailable lysine acetyltransferase 2A (KAT2A) and lysine acetyltransferase 2B (KAT2B) degrader, in participants with relapsed/refractory acute myeloid leukemia (AML) or myelodysplastic syndromes (MDS). The study consists of two parts: Part A (Dose Escalation) to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D), and Part B (Dose Optimization) to further evaluate safety, PK, PD and efficacy at selected dosages.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant must be ≥18 years of age
2. Participant must have confirmed diagnosis as follows:

   R/R AML and has not achieved adequate response to, cannot tolerate, or refused all approved therapies known to be active for treatment of their disease OR R/R MDS with over 10% blasts in the bone marrow and has not achieved an adequate response to at least 4 cycles of a hypomethylating agent (HMA)- containing regimen or other treatment known to be active for their disease OR R/R AML or R/R MDS that has relapsed after a hematopoietic stem cell transplant (HSCT)
3. Participant must be willing and able to comply with scheduled study visits and treatment plans.
4. Participant must be willing to undergo all study procedures unless contraindicated due to medical risk.
5. Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤2
6. Participant must have adequate hepatic function
7. Participant must have adequate renal function
8. Participant must have adequate cardiovascular function
9. Participant must have a white blood cell (WBC) count ≤20 × 10⁹/L (with stable hydroxyurea use allowed)
10. Participant must meet timing requirements with respect to prior therapy and surgery
11. Participant must agree to use effective contraception during the study and for the required post-treatment period: Males: Use condoms (even if vasectomized) during the study and for 90 days post-treatment. Females of childbearing potential: Use a combination of 1 highly effective and 1 effective method of contraception during the study and for 180 days post-treatment.

Key Exclusion Criteria:

1. Participant is unable to provide informed consent and/or to follow protocol requirements.
2. Participant has undergone chimeric antigen receptor T cell therapy or HSCT within 60 days of the first dose of study treatment or has active clinically significant graft-versus-host disease (GVHD)
3. Participant has another malignancy that may interfere with diagnosis and treatment of R/R AML or R/R MDS.
4. Participant has an active severe infection that requires anti-infective therapy or has an unexplained temperature of >38.5°C during screening visits or on their first day of study treatment.
5. Participant has a known sensitivity to AUTX-703 or any of its components.
6. Participant is taking systemic strong CYP3A4 inhibitors or inducers within 14 days of the first dose of study treatment.
7. Participant who are taking proton pump inhibitors should be switched to another acid-reducing agent such as an antacid or H2 blocker
8. Participant is taking P-gp and breast cancer resistance protein (BCRP) inhibitors or inducers within 14 days of first dose of study treatment.
9. Participant has active hepatitis B virus (HBV) or hepatitis C virus (HCV) infections with detectable viral load
10. Participant has experienced AIDS related illness within the past 6 months or have detectable HIV viral load.
11. Participant has an uncontrolled intercurrent illness
12. Participant has active Class III or IV cardiovascular disease within 6 months prior to the start of study treatment
13. Participant is unable to tolerate the administration of oral medication or has GI dysfunction that would preclude adequate absorption, distribution, metabolism, or excretion of an oral medication
14. Participant is pregnant or breastfeeding or is planning to become pregnant within 1 year of the start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs), Dose-Limiting Toxicities (DLTs), and Serious Adverse Events (SAEs) | From the first dose through 28 days after the last dose of study drug.
  To assess the safety and tolerability of AUTX-703 by evaluating the incidence and severity of AEs, DLTs, SAEs, and AEs leading to treatment discontinuation.

SECONDARY OUTCOMES:
To Identify the Recommended Phase 2 Dose (RP2D) of AUTX-703 | From the first dose through 28 days after the last dose of study drug.
  To determine the RP2D of AUTX-703 based on safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary clinical activity data.
Peak Plasma Concentration (Cmax) | From the first dose through the first treatment cycle (28 days)
Time to Maximum Concentration (Tmax) | From the first dose through the first treatment cycle (28 days)
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinity (AUCinf) | From the first dose through the first treatment cycle (28 days)
Area Under the Plasma Concentration-Time Curve to the Last Measurable Concentration (AUClast) | From the first dose through the first treatment cycle (28 days)
Elimination Half-Life (t½) | From the first dose through the first treatment cycle (28 days)
Apparent Clearance (CL/F) | From the first dose through the first treatment cycle (28 days)
Apparent Volume of Distribution (Vd/F) | From the first dose through the first treatment cycle (28 days)
To characterize the PD of AUTX-703 | From the first dose through 28 days after the last dose of study drug
  To evaluate changes in KAT2A and KAT2B levels in peripheral blood and bone marrow as markers of pharmacodynamic response
AML: Complete remission (CR) rate | Up to 18 months
AML: CR + CRh rate | Up to 18 months
AML: Duration of CR | Up to 18 months
AML: Duration of CR + CRh | Up to 18 months
Objective response rate (ORR) | Up to 24 months
AML: Duration of response (DOR) | Up to 18 months
AML: Transfusion independence (TI) rate | Up to 18 months
AML: Event free survival (EFS) | Up to 24 months
AML: Overall survival (OS) | Up to 24 months
MDS: Complete remission (CR) rate | Up to 18 months
MDS: PR rate | Up to 18 months
MDS: CR+PR rate | Up to 18 months
MDS: Duration of CR | Up to 18 months
MDS: Duration of PR | Up to 18 months
MDS: Duration of CR+PR | Up to 18 months
MDS: Event free survival (EFS) | Up to 24 months
MDS: Overall survival (OS) | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - City of Hope National Medical Center, Duarte, California
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Ohio State University, The James Comprehensive Cancer, Columbus, Ohio
  - UPENN Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Sarah Cannon Center for Blood Cancer at TriStar Centennia, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas